CLINICAL TRIAL: NCT04509297
Title: Effects of High-protein Milk Supplementation on Muscular Strength and Power, Body Composition, and Skeletal Muscle Regulatory Markers Following Heavy Resistance Training in Resistance-trained Men
Brief Title: Resistance Training and Milk Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marymount University (Other)
Collaborators: University of Tehran (Other)
Responsible Party: Principal Investigator, Alexei Wong, Assistant Professor, Marymount University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Sports sciences institute.1396
Record Dates: First submitted 2020-08-05; First posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Muscular Hypertrophy
Keywords: Hypertrophy; body composition; milk; resistance training
MeSH Terms: conditions — Hypertrophy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High protein milk (Experimental): Experimental: High protein milk consumption This arm involved High protein milk whole consumption concomitant with 6 weeks of resistance training. Subject ingested consumed 1 x 250 mL immediately after resistance training and 1 x 250 mL half an hour before bedtime.
  Interventions: Dietary Supplement: high protein milk; Dietary Supplement: Placebo
- Placebo (Placebo Comparator): This arm involved consumption of a maltodextrin drink with a 9% solution with a vanilla flavor concomitant with 6 weeks of resistance training. Subject ingested consumed 1 x 250 mL immediately after resistance training and 1 x 250 mL half an hour before bedtime. drink r
  Interventions: Dietary Supplement: high protein milk; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: high protein milk — This intervention consisted of high protein milk consumption concomitant with 6 weeks of resistance training. Subject ingested consumed 1 x 250 mL immediately after resistance training and 1 x 250 mL half an hour before bedtime.
Dietary Supplement: Placebo — This intervention consisted of the consumption of a maltodextrin drink with a 9% solution with a vanilla flavor concomitant with 6 weeks of resistance training. Subject ingested consumed 1 x 250 mL immediately after resistance training and 1 x 250 mL half an hour before bedtime.

SUMMARY:
Post-resistance training high protein milk supplementation may be a viable method to elicit muscular gains.

The investigators hypothesis is that high protein milk supplementation would improve skeletal regulatory markers, hormonal responses and body composition in resistance-trained men.

DETAILED DESCRIPTION:
The aim of this investigation was to compare the effects of high protein milk supplementation (daily and after training sessions) during 6 weeks of resistance training on skeletal muscle regulatory markers, hormonal responses and body composition in resistance-trained men. Specific aims of the study are to:

To investigate the extent to which high protein milk supplementation will improve anabolic factors, lean body mass, fat mass and decrease catabolic markers after 6 weeks of resistance training in resistance-trained men.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-35 years of age
* Healthy Males
* Experienced at resistance training (at least 1 year of prior structured resistance training 3 x week).

Exclusion Criteria:

* smoking
* chronic alcohol consumption
* having any medical issues and diseases
* lactose intolerance
* the consumption of any dietary supplements (including vitamins or protein supplements) or medications for 6 months prior to participation

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2018-05-05 (Actual); Study Completion 2018-05-05 (Actual)

PRIMARY OUTCOMES:
Circulatory Myokines levels | 6 weeks
  Fasting blood samples were collected from the antecubital vein using standard procedures and then analyzed to establish concentration of myostatin and follistatin.
Circulatory hormone levels | 6 weeks
  Fasting blood samples were collected from the antecubital vein using standard procedures and then analyzed to establish concentrations of testosterone, IGF-1, growth hormone, insulin and cortisol
Body composition | 6 weeks
  Lean body mass and body fatness will be evaluated using bioelectrical impedance

SECONDARY OUTCOMES:
Muscular Strength | 6 weeks
  Using a 1 repetition maximum test (defined as the maximal weight an individual can lift for only one repetition) for the bench press and back squat exercises
Muscular Power | 6 weeks
  Using the Wingate test

CONTACTS AND LOCATIONS:
Overall Officials: Alexei Wong, Principal Investigator — Marymount University
Locations (1):
- Marymount University, Arlington, Virginia, United States

IPD SHARING:
Plan to Share IPD: No